CLINICAL TRIAL: NCT05851144
Title: South Texas Early Prevention Studies SNAP-Ed
Brief Title: South Texas Early Prevention Studies SNAP-Ed (STEPS SNAP-Ed)
Acronym: STEPSSNAP-Ed
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Rio Grande Valley (Other)
Collaborators: Health and Human Services Commission (HHSC) (Unknown); Pharr-San Juan-Alamo Independent School District (Unknown); La Joya Independent School District (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STEPS SNAP-Ed
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Health-Related Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: School-based approach is used to complete the randomized assignment to intervention or control conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention arm involves participants to the Bienestar/Neema Coordinated School Health Program (BN CSHP), a Texas Education Agency-approved school health curricula with multi-prong interventions.
  Interventions: Behavioral: Bienestar/Neema Coordinated School Health Program (BN CSHP)
- Control (No Intervention): Participants in the control group follow regular routine with physical activities, food service, and parental engagment.

INTERVENTIONS:
Behavioral: Bienestar/Neema Coordinated School Health Program (BN CSHP) — Bienestar/Neema Coordinated School Health Program (BN CSHP), a Texas Education Agency-approved school health curricula, is a multi-prong intervention
  Arms: Intervention

SUMMARY:
The "South Texas Early Prevention Studies Supplemental Nutrition Assistance Program-Education" (STEPS SNAP-Ed) is a project designed to control and prevent obesity rates in South Texas children. The University of Texas Rio Grande Valley (UTRGV) was awarded funding from the Texas Health and Human Services Commission (HHSC) to provide behaviorally focused, evidence-based nutrition education and obesity prevention interventions to serve the South Texas SNAP-Ed target audience. The SNAP-Ed target audience are SNAP-Ed recipients, SNAP eligible, communities with ≥50% low-income, schools where ≥50% of children are on free and reduced meals, and those on Medicaid. Specifically, the STEPS SNAP-Ed Project will engage parents, school staff, hospital staff and community members to make healthier food choices available and encourage physical activity to control and prevent obesity in preschool children. The STEPS SNAP-Ed Project is a collaborative effort among a university, two school districts, and a hospital system in the Rio Grande Valley.

DETAILED DESCRIPTION:
The STEPS SNAP-Ed project aim is to meet the United States Department of Agriculture's (USDA) Food and Nutrition Service (FNS) requirements through the following Texas SNAP-Ed State Goals:

State Goal I: Implement health promotion activities to help the SNAP-Ed Target Audience establishes healthy eating habits and a physically active lifestyle. State Goal II: Reduce risk factors for chronic diseases such as obesity, type 2 diabetes, and cardiovascular disease among the SNAP-Ed Target Audience. State Goal III: Increase partnership collaboration of nutrition, physical activity, and wellness education across the state.

State Goal IV: Increase consumption of fruits, vegetables, and other foods that comprise a healthy diet among the SNAP-Ed Target Audience in accordance with Dietary Guidelines for Americans 2015-2020 8th Edition.

State Goal V: Increase ongoing physical activity among the SNAP-Ed Target Audience in accordance with Physical Activity Guidelines 2nd Edition. State Goal VI: Increase Policy, Systems, and Environmental (PSE) projects consistent with Fiscal Year 2021 SNAP-Ed Plan Guidance.

Specifically, the primary and secondary outcomes are the following:

II.a. Primary Outcome - Obesity Prevalence

1) Decrease obesity prevalence by 5 percent in children from intervention schools compared to those in control schools over the 3-year intervention period.

II.b. Secondary Outcomes - Fitness and Dietary Intake

1. Significantly increase fitness scores of children in intervention schools compared to those in control schools over the 3-year intervention period.
2. Significantly increase the intake of fruits, vegetables, and whole grains servings in children from intervention schools compared to those in control schools over the 3-year intervention period.

II.c. Evaluation Plan - Summary

1. BMI Measure. Obesity prevalence is measured by height (ht.), weight (wt.) and body mass index (BMI) calculated by (kg/m2). Obesity prevalence is defined by a BMI ≥ 95th percentile.
2. Fitness Measure. Fitness test consists of the modified PACER test (15-meter distance, 20-meter cadence). It is modified because the PACER fitness test was designed to begin implementation in third grade. The PACER test involves running back and forth across a course to a cadence audio track played from a CD. Beeps in the track indicate when a child should reach the end point of a lap. The fitness test begins at a slow pace and it gets more difficult as the pace quickens. The child continues running until he/she fails to complete a lap by reaching the end point before the next beep on the meter cadence track. Once a child misses two laps (missed laps do not need to be consecutive) the PACER Test concludes, and the number of laps is recorded.
3. Dietary Intake Measure. Dietary Intake of fruits, vegetables, and whole grains consumed during school breakfast and lunch will be measured by direct observation and supplemented by meal photographs (before and after meals are consumed). Dietary data will be collected over 3 consecutive days and consumption average will be calculated.
4. Process Evaluation Measures.

   1. Dose (lesson plan taught) & reach (number of participants in attendance) and submitted into PEARS software.
   2. SNAP Ed long-term, mid-term and short-term survey instruments will be submitted into PEARS software.

ELIGIBILITY:
Inclusion Criteria:

* All enrolled PreK 4 students to participating school districts

Exclusion Criteria:

* None

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1104 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
A rate of 5% decrease in BMI | 3 years
  Number of participants in the intervention schools, as compared to the control schools, will demonstrate a 5% decrease at the rate of childhood obesity as measured by the BMI>=95 Percentile

SECONDARY OUTCOMES:
Fruits/vegetables/whole grains consumption increase at a rate of 5% increase in servings | 3 years
  The number of fruits/vegetables/whole grains consumption increase in servings at a rate of 5%
A rate of 5% Increase of pacer laps run as measured by laps recorded | 3 years
  A rate of 5% Increase of pacer laps run as measured by laps recorded

CONTACTS AND LOCATIONS:
Overall Officials: Zasha Romero, Ph.D., Principal Investigator — University of Texas Rio Grande Valley
Locations (1):
- University of Texas Rio Grande Valley, Edinburg, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregated data will be shared.

DOCUMENTS (1):
  • Informed Consent Form (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT05851144/ICF_000.pdf